CLINICAL TRIAL: NCT06080932
Title: Ketogenic Intervention in Depression
Acronym: KIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022H0271
Record Dates: First submitted 2023-06-01; First posted 2023-10-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Depression; Ketosis
MeSH Terms: conditions — Depression; Ketosis | interventions — Diet, Ketogenic; Blood Specimen Collection; Ketones; Body Composition; Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketogenic Diet (Experimental): The KD will follow general principles as we have described with the aim to achieve blood ketones >0.5 mM, which will require most participants to consume <50 g/day carbohydrate and ~1.5 g/kg reference weight protein. Fat will comprise the remaining calories with an emphasis on monounsaturated and saturated sources from whole foods.
  Interventions: Other: Ketogenic Diet; Other: NIH Toolbox; Other: gradCPT; Other: Resting-state fMRI; Other: Task-fMRI; Other: CGM/CKM; Biological: Blood Draw; Other: Sleep Monitoring; Biological: Ketone/Glucose Monitoring; Other: Body Composition; Behavioral: PHQ-9; Behavioral: WHO-5; Behavioral: SKID

INTERVENTIONS:
Other: Ketogenic Diet — The diet intervention will start after all baseline testing is complete
Other: NIH Toolbox — IPAD-based assessments that examines cognitive function
Other: gradCPT — The gradCPT contains grayscale photographs of mountain scenes and city scenes. Scene images gradually transition from one image to the next
Other: Resting-state fMRI — Whole brain echo-planar imaging (EPI) volumes sensitive to the BOLD signal will be acquired. Images will be re-aligned, un-warped, and normalized. Confounding effects of white matter, CSF signal, and head motion will be regressed from the functional time series, followed by bandpass filtering, linear detrending and smoothing, and whole brain resting state networks will be identified (e.g., default mode network, salience network, etc).
Other: Task-fMRI — During whole brain EPI data acquisition, participants will be presented with words and pictures and asked to make judgements about the stimuli, such as indicating whether a particular stimulus (e.g., face-name association, word, number, or letter) has been previously presented, if a presented stimulus is a city or mountain scene, the direction an arrow is pointing (left or right), if a pair of stimuli match (e.g., faces with neutral or emotional expressions; word with a face). Behavioral responses will be recorded with an MRI compatible button box.
Other: CGM/CKM — Continuous Ketone/Glucose Monitor will be applied at the start of Test Day 1. The sensor will be checked by the study team at each test day and will be removed and replaced by a fresh sensor at ~2- week intervals during the study. The sensor will be removed at the end of the final test day.
Biological: Blood Draw — Blood samples will be collected according to the schedule in Figure 1
Other: Sleep Monitoring — Sleep will be assessed by ring-based acceleration with cloud technology (Oura Ring). This monitor is less burdensome than other sleep monitoring technologies and less likely to interfere with normal sleep and activity demands. Worn daily throughout intervention
Biological: Ketone/Glucose Monitoring — KetoMojo hand-held glucometer will be used daily to monitor dietary intervention adherence.
Other: Body Composition — DEXA Scanning will be done pre-, mid-, and post- intervention.
Behavioral: PHQ-9 — It is a self-assessment tool used to screen and assess the severity of depression in individuals. The PHQ-9 consists of nine questions based on the nine criteria for diagnosing major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
Behavioral: WHO-5 — The WHO-5, also known as the World Health Organization-Five Well-Being Index, is a self-assessment tool used to measure subjective well-being and mental health. It was developed by the World Health Organization (WHO) as a brief and reliable instrument to evaluate well-being in clinical and research settings.
Behavioral: SKID — The SKID refers to the Structured Clinical Interview for DSM Disorders (SCID). It is a widely used diagnostic tool in the field of psychiatry and clinical psychology. The SCID is a semi-structured interview designed to assess and diagnose various mental disorders according to the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM), which is published by the American Psychiatric Association.

SUMMARY:
The goal of this study is to examine whether a well-formulated ketogenic diet (KD) can be implemented into a university counseling treatment program for major depression and to test whether such a program has any benefit on mental and metabolic health.

DETAILED DESCRIPTION:
Major depression is a burgeoning problem that affects over five percent of adults worldwide and is rapidly increasing in the United States. From the second quarter of 2019 to June of 2020, the prevalence of symptoms of depression spiked from 6.5 to 24.3% , which was largely attributed to the COVID-19 pandemic. Major depression and suicidal ideation have increased markedly in young adults, particularly within college campuses. In 2020, counselors at the Ohio State University (OSU) experienced a surge in the number of students with various mental health issues with anxiety and depressive disorders being the most common. The escalating prevalence of depression bubbling under the surface of the ongoing COVID-19 pandemic represents a unique challenge that requires new and creative solutions.

Recently, a KD was administered to adults who had been admitted to a psychiatric hospital and were suffering from various mental disorders. The dietary intervention lasted between 16 and 248 days and showed significant improvements in depression and psychotic symptoms. Ketogenic diet interventions (and ingestion of ketone esters) have also been associated with more stable brain networks, assess with functional Magnetic Resonance Imaging (fMRI). Additionally, a novel but as yet under-appreciated effect of nutritional ketosis is to induce a broad-spectrum reduction in inflammation in metabolically-impaired individuals. Elevations in a range of inflammation biomarkers has been associated with severity of depression.

Although KDs have been proposed as a treatment option for mental health disorders, including schizophrenia and depression, few human clinical trials have tested the efficacy of this eating pattern specifically in a population of adults with major depression. In patients with type 2 diabetes (n=262) prescribed a KD using a novel virtual care model (Virta Health), we observed significant improvements in depressive symptoms after 10-weeks, which were directly correlated with the degree of carbohydrate restriction and nutritional ketosis as assessed by blood concentrations of ketones.

ELIGIBILITY:
Inclusion Criteria:

* OSU students (age 18-30 years at the time of enrollment) with confirmed major depressive disorder as determined by SCID-5 diagnosis at baseline testing.
* Currently engaged in counseling treatment for depression at CCS
* Available for a 12-week period and indicate willingness and ability to eat KD foods as prescribed

Exclusion Criteria:

* Disordered eating, as evidenced by meeting criteria for Anorexia Nervosa, Bulimia Nervosa, Binge Eating Disorder, Other Specified Eating Disorder, Unspecified Eating Disorder, or Avoidant Restrictive Eating Disorder during the SCID-5 interview at baseline testing.
* Substantial imminent risk of suicide as assessed during the SCID-5 interview.
* Body mass index (BMI) < 20 kg/m2
* Habitual consumption of a structured low-carbohydrate diet in the last 6-months
* Gastrointestinal disorders or allergies that would prevent adherence to prescribed diets
* Alcohol consumption in excess of 3 drinks/daily or 14 drinks/weekly
* Diagnosed diabetes, liver, kidney, or other metabolic or endocrine dysfunction, or use of diabetic medications other than metformin
* Inability to access or prepare appropriate KD foods/meals
* Pregnant, lactating, or planning on becoming pregnant during the study
* Unwilling to perform finger-stick blood testing or continuous glucose/ketone monitoring

Exclusion for optional MRI:

• The CCBBI screening form (https://redcap.osumc.edu/redcap/surveys/?s=N3XJ4WC7T9) will be used to assess MRI eligibility. Endorsement of items that contraindicate MRI will serve as exclusion criteria (pacemaker, stint, claustrophobia, etc.).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
WHO-5 Questionnaire | Up to ~ 12 weeks
  The WHO-5 (World Health Organization-Five Well-Being Index) is a self-assessment questionnaire used to measure subjective well-being and mental health. It was developed by the World Health Organization (WHO) and consists of five statements related to positive mood, vitality, and general interest in life. The five statements in the WHO-5 questionnaire are as follows:
  I have felt cheerful and in good spirits. I have felt calm and relaxed. I have felt active and vigorous. I woke up feeling fresh and rested. My daily life has been filled with things that interest me. Respondents are asked to rate each statement based on how they have felt over the past two weeks, using a six-point Likert scale ranging from "at no time" to "all of the time." The scores for each item are summed, resulting in a total score ranging from 0 to 25. Higher scores indicate better well-being
The Hamilton Depression Scale | Up to ~ 12 Weeks
  Hamilton Depression Scale consists of 17 items that cover various symptoms of depression, including depressed mood, guilt, suicidal thoughts, insomnia, agitation, weight loss, and somatic symptoms. Each item is rated on a scale from 0 to 4 or 0 to 2, depending on the item, with higher scores indicating more severe symptoms.
  The scale is typically administered by a trained healthcare professional who interviews the individual and rates their symptoms based on their observations and the individual's self-report. The rater assesses the severity of each symptom and determines the appropriate score for each item.
  The total score on the Hamilton Depression Scale can range from 0 to 52, with higher scores indicating greater severity of depression. However, it is important to note that the interpretation of the total score requires clinical judgment and consideration of the individual's overall presentation and context.
Finger Stick BHB | Up to ~ 12 Weeks
  changes in fasting ketone levels.
Finger Stick Glucose | Up to ~ 12 Weeks
  changes in fasting glucose levels.

SECONDARY OUTCOMES:
PHQ-9 | Up to ~ 12 Weeks
  The Patient Health Questionnaire-9 used bi-weekly to asses changes in degree of depression (intensity and severity).
  Each item in the PHQ-9 is rated on a scale from 0 to 3, reflecting the frequency of the symptoms over the past two weeks. The response options are "not at all" (0), "several days" (1), "more than half the days" (2), and "nearly every day" (3). The scores for each item are summed to obtain a total score ranging from 0 to 27.
  The interpretation of PHQ-9 scores is as follows:
  0-4: None to minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20 and above: Severe depression
CGM/CKM | Up to ~ 12 Weeks
  changes in daily glucose and ketone levels.
Metabolic Panel | Up to ~ 12 Weeks
  Changes in metabolic blood panel will be assessed at in lab visits (eg. Baseline, Week 6, and Week 12)
Blood Pressure | Up to ~ 12 Weeks
  Changes in both Systolic and Diastolic blood pressure will be measured at each lab visit (eg. Baseline, Week 6, and Week 12).
  Recording: The systolic and diastolic pressures are recorded in millimeters of mercury (mmHg). For example, a reading of "120/80 mmHg" indicates a systolic pressure of 120 mmHg and a diastolic pressure of 80 mmHg.
Cognitive Testing | Up to ~ 12 Weeks
  The NIH Toolbox includes a comprehensive set of measures across various domains, including:
  Cognition: executive function, attention, memory, language, processing speed, and working memory. These measures help evaluate cognitive abilities and identify potential cognitive impairments.
  Emotion: emotional well-being, social functioning, and psychological distress. It provides tools to assess symptoms of depression, anxiety, and positive affect, as well as social functioning and quality of life.
  Motor: motor function, dexterity, strength, coordination, and balance. These assessments are designed to evaluate both fine and gross motor skills and detect any motor impairments or changes over time.
  Sensation: auditory, visual, and somatosensory abilities. These measures help evaluate sensory perception, discrimination, and thresholds.
Task-fMRI | Up to ~ 12 Weeks
  During whole brain EPI data acquisition, participants will be presented with words and pictures and asked to make judgements about the stimuli, such as indicating whether a particular stimulus (e.g., face-name association, word, number, or letter) has been previously presented, if a presented stimulus is a city or mountain scene, the direction an arrow is pointing (left or right), if a pair of stimuli match (e.g., faces with neutral or emotional expressions; word with a face). Behavioral responses will be recorded with an MRI compatible button box.
Resting State fMRI | Up to ~ 12 Weeks
  Changes in cortical thickness, brain volume, and functional connectivity for pre- intervention and post intervention testing days.
  Whole brain echo-planar imaging (EPI) volumes sensitive to the BOLD signal will be acquired. Images will be re-aligned, un-warped, and normalized. Confounding effects of white matter, CSF signal, and head motion will be regressed from the functional time series, followed by bandpass filtering, linear detrending and smoothing, and whole brain resting state networks will be identified (e.g., default mode network, salience network, etc).
Lean Body Mass (kg) | Up to ~ 12 Weeks
  Changes in lean body mass.
Changes in BMI | Up to ~ 12 Weeks
  Changes in body mass index.
Changes in total body weight ( kg) | Up to ~ 12 Weeks
  Changes in total body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06080932/Prot_000.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06080932/ICF_001.pdf